CLINICAL TRIAL: NCT00125580
Title: Healthy Sleeping and Feeding During Infancy: Pilot Study for the Primary Prevention of Obesity in Primary Care
Brief Title: Healthy Sleeping and Feeding During Infancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20970EP
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Obesity
Keywords: Obesity; Childhood Obesity; Infant Sleep; Infant growth; Infant feeding
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Behavioral: Infant sleep instruction

SUMMARY:
Childhood obesity has reached epidemic proportions and its prevalence continues to rise, even among very young children. A recent report from the National Health and Nutrition Examination Survey (NHANES) revealed that from 1999 to 2002, 10.3% of children ages 2 to 5 were overweight, an increase from 7% in 1994. Epidemiologic evidence is now emerging that suggests obesity in childhood and adulthood may often originate from accelerated weight gain during infancy. Further data are accumulating that link short sleep duration with obesity during childhood and later life. Prospective data are lacking that demonstrate whether the accelerated weight gain during infancy can be prevented and whether interventions to improve sleep early in life can prevent childhood obesity.

Key Objectives:

The key objectives are:

* To adapt a procedure aimed at prolonging sleep duration during infancy that is effective in experimental settings to the clinical setting of primary care; and
* To evaluate, in the primary care setting, the effect of a simple training procedure on overnight sleep duration and rate of weight gain during the first four months of life.

DETAILED DESCRIPTION:
The objective of this proposal is to test, in a primary care setting, the effect of an established intervention designed to promote healthy feeding and sleeping behaviors early in life on risk factors for subsequent obesity. Because nocturnal feeding of infants, short sleep duration, and childhood obesity are linked, the procedure is designed to prevent short sleep duration and subsequently accelerated weight gain during infancy, two emerging risk factors for obesity in childhood and adulthood. In this study, 40 participants will be randomized to receive either an intervention that teaches infants to sleep through the night by 8 weeks of age or standard care. The procedure instructs parents to offer a "focal feed" before bedtime, avoid feeding as the first alternative to infant waking and distress, and carry out environmental control measures that emphasize day/night differences. In assessing the impact of the intervention, night wakening, and rate of weight gain will be assessed between birth and 4 months of age. The current proposal will test the feasibility of delivering this proven intervention in the primary care setting, an environment that must be included in primary preventive strategies for childhood obesity.

Aim 1: To adapt a procedure aimed at prolonging sleep duration during infancy that is effective in experimental settings to the clinical setting of primary care.

This procedure, which instructs parents to offer a "focal feed" before bedtime, avoid feeding as the first alternative to infant waking and distress, and carry out environmental control measures that emphasize day/night differences has been successful at prolonging sleep duration in experimental settings. By demonstrating that subjects can be recruited from the newborn nursery, be taught the procedure at a primary care visit, and followed for four months, the feasibility of a larger study will be more apparent to external funding agencies.

Aim 2: To evaluate, in the primary care setting, the effect of a simple training procedure on overnight sleep duration and rate of weight gain during the first four months of life.

It is hypothesized that the positive effect of the procedure in an experimental setting will be replicated in a randomized controlled trial in the primary care setting. By definition, teaching infants to sleep through the night will be manifest in longer sleep duration, which has been shown to be protective for childhood obesity in epidemiological studies. Sleeping through the night is hypothesized to promote protective factors for childhood obesity by supporting

ELIGIBILITY:
Inclusion Criteria:

* ≥37 weeks gestation
* Primiparous mother (first pregnancy)
* Singleton
* Breast or bottle-fed
* Birth weight ≥2500 grams

Exclusion Criteria:

* <37 weeks gestation
* Multiparous mother {see above comment}
* Twin or multiple infant
* Birth weight <2500 grams
* Maternal conditions causing prolonged hospital stay or "non-routine" postpartum follow-up (except for diabetes mellitus: type 1, 2, or gestational)
* Infants with chronic illnesses or anomalies that require non-routine care or follow-up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The rate of sleeping through the night at 8 weeks of age between treatment groups (intervention versus standard treatment)

SECONDARY OUTCOMES:
Across the study period, infant weight gain will be measured to study differences between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Paul, MD, MSc, Principal Investigator — Milton S. Hershey Medical Center
Locations (2):
- United States (2):
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State University, University Park, Pennsylvania